CLINICAL TRIAL: NCT06509776
Title: Early Life Determinants of Skeletal Maturation and Endocrine Health in Young Adults - A Nationwide Birth Cohort Study
Brief Title: Skeletal Maturation and Endocrine Health in Young Adults
Acronym: EPIPEAK
Status: Enrolling by invitation | Type: Observational
Sponsor: Holbaek Sygehus (Other)
Collaborators: Aarhus University Hospital (Other); Aalborg University Hospital (Other); University of Southern Denmark (Other); University Hospital Bispebjerg and Frederiksberg (Other); Zealand University Hospital (Other); Odense University Hospital (Other); Rigshospitalet, Denmark (Other); Statens Serum Institut (Other); Hvidovre University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: S-20230105; NNF22OC0080437 (Other Grant/Funding Number: Novo Nordisk Foundation); 21-B-0436 (Other Grant/Funding Number: Helsefonden, Denmark)
Record Dates: First submitted 2024-07-15; First posted 2024-07-19 (Actual); Last update posted 2025-01-10 (Actual); Status verified 2025-01

CONDITIONS: Osteoporosis; Sarcopenia; Obesity; Cardiovascular Diseases
Keywords: Bone and Bones; Bone mineralization; Bone mineral density; Bone density; Endocrinology; Hormones; Thyroid Hormones; Parathyroid Hormone; Puberty; Adolescent; Glucocorticoids; Genetics; Human Genetics; Epigenomics; Neonatal Screening; Body Composition; Cohort Study; Epidemiology; Phenotype
MeSH Terms: conditions — Osteoporosis; Sarcopenia; Obesity; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood will be drawn for plasma analyses for endocrine status and biomarkers of bone metabolism (outcomes). Hair samples will be collected for cortisol (outcomes). Already collected neonatal blood samples will be measured for genetic and epigenetic profiles (predictors).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Population sample: Random subsample of all 17-18-year-old individuals in Denmark, i.e. live births from year 2006 and 2007.

SUMMARY:
Diseases which can be the result of poor lifestyle choices in adult life, such as osteoporosis, obesity or poor muscle mass (sarcopenia) can also be driven by heritable genetic factors. More surprisingly, perhaps, the genes we inherit from our parents can be modified as a result of influences that affected the health and pregnancy of our mothers and hence the environment experienced in the womb and at birth. The purpose of this study is to investigate which factors are needed for good bone health and hormonal health in young adulthood as well as good muscle mass and normal fat mass, and how this is influenced by factors before birth and by childhood health. Specifically, we will measure bone mass and body composition in young adults (18 years of age) and measure hormones in blood and in hair samples. The clinical visits will be available nationwide at several centers to make participation swift and easy for participants. The changes (known as epigenetic modification) to genes at birth will be studied in dried blood spot samples stored from birth 18 years ago in the Danish Serum Institute and we will use national health registers to identify factors during pregnancy and in childhood that contribute to health effects at age 18.

DETAILED DESCRIPTION:
Population-based, nationwide, cross-sectional, clinical study with already available early life exposure data including bio banked neonatal biological samples. An embedded design using the full 2006+2007 birth cohorts is used to demonstrate external validity of the clinically assessed cohort. We will obtain the necessary ethics and regulatory approval and individual consent from the participants who are all aged 18.

The overall aim of the project addresses whether the following sets of potential determinants are associated with young adult hormonal status, lipids, bone turnover markers, bone mineral density (BMD), fat mass and lean body mass at age 18 years: a) maternal risk factors during preconception and pregnancy; b) risk factors at birth; c) neonatal epigenetic signature; d) childhood risk factors.

Aim 1 - Epigenetics - Is peak bone mass and body size influenced by epigenetic profile for endocrine signals at birth? From the second trimester of pregnancy and until early adulthood, bone is gradually developed and shaped, with longitudinal growth dominating the later stages of fetal life, infancy, and childhood. This is followed by a period of rapid bone mineral accrual occurring up to and during puberty, with bone mass accretion ultimately reaching a plateau in young adult life. It is strongly suggested by prior research that epigenetic variation at birth can result from differences in maternal health, lifestyle, nutrition, smoking and medication usage and result in long-term changes in gene expression and metabolism.

As existing childhood cohorts either lack BMD information, suffer from significant cohort attrition, and low recruitment success, there is an opportunity to instead use national invitations to recruit directly into an efficient endocrine and bone outcomes study and use already archived biological material from early infancy and register data and obtain individual study subject consent.

Aim 2 - Endocrine status in young adulthood - Does maternal medication use and health issues prior to pregnancy or in pregnancy affect endocrine health in young adults? This question will be addressed using data from Danish national registers. While it is straightforward to link binary events data e.g., malformations or paediatric admissions (eg epilepsy, diabetes, failure to thrive) to registry capture of their maternal exposures, we will be obtaining detailed information about continuous outcomes including endocrine serum biochemistry (thyroid axis, GH axis, PTH-vitamin D-calcium axis, lipids, HbA1c), hair cortisol levels (a cumulative serum cortisol metric) as well as body composition and bone density metrics.

Aim 3 - DXA measured muscle, fat mass and lipid status in young adults - Do suboptimal conditions prior to pregnancy, during pregnancy, birth, and childhood, such as lifestyle, poor health and low socioeconomics adversely influence establishment of healthy body composition and lipid status in young adulthood? Detailed register-based information prior to pregnancy, about pregnancy, birth and childhood health will be used to identify areas open to prevention. Detailed information will be obtained via the Danish national health registers.

Statistical consideration - With a study population of 2,000, the power (given α=0.05) available to detect a 0.2 SD effect on a continuous outcome such as PBM for a risk factor with a population prevalence of 20% is 90%. With inclusion of 1,500 subjects, the corresponding study power is 90% for detection of an effect size of 0.24 SD or 80% for detection of an effect size of 0.2 SD. The study needs this resolving power to be able to address multiple contributing factors and for the inclusion of factors in the model that may have a population prevalence below 20%. Less common factors would, even if powerful drivers of skeletal health, be somewhat less useful in population impact even if successfully modified.

Biological material - All material for use in the current project will be stored in a research biobank during the current study during its term. Any remaining material is transferred to biobank for future research with the approval of the Danish Data Protection Agency. The purpose of the biobank is to ensure validation of the analysis methods used over time. The participants must give consent to the storage of their biological material in the biobank. It is completely optional if the participants want to donate their excess biological material to the biobank and if they do not want this, it does not affect their participation in the study. For new research, new consent must be obtained, but the Scientific Ethics Committee can grant exemption from the consent requirement.

All material will be stored in compliance with Danish legislation on data protection.

24 mL of blood will be drawn. All blood samples are encoded so that all samples are anonymized, and the key is under special protection and only with access for authorized personnel. All extra material will be kept in the biobank.

To ensure uniformity between neonatal and adolescent samples, DBS will be created from the freshly drawn whole blood. DBS are created by spotting 3x75µL onto a cotton filter paper of the same type used in 2006-2007. The cards are left overnight at ambient temperatures then transferred to -20C for long term storage. DNA is be extracted from two 3.2mm disks excised from the DBS card, then purified using magnetic silica beads. Finally, concentrations are measured using intercalating dyes.

All hair samples (minimum 20 mg per participant) will be encoded so that all samples are pseudonymised, and the key is under special protection and only with access for authorized personnel. All hair samples will be used in the analyses, and then discarded.

ELIGIBILITY:
Inclusion Criteria:

* Individuals (n = 2000) born in Denmark in 2006 or 2007
* Are 18 years old and alive at the time of the clinical examination

Exclusion Criteria:

* Pregnancy or lactation
* No DBS samples available
* Lack of consent to use DBS samples or national health registries
* Emigration or disappearance

Ages: 18 Years to 19 Years | Sex: All
Age Groups: Adult
Study Population: The Danish Personal Civil Registration will be used to identify all alive individuals born in Denmark in 2006 and 2007 using civil registration numbers. Invitations will be sent through secure e-mail (E-boks) in blocks until 2,000 participants have been reached. The study population will be selected with representative geographical distribution in Denmark.
Sampling Method: Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2024-11-11 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2031-09 (Estimated)

PRIMARY OUTCOMES:
Bone Mineral Density of Spine, Hip and Whole-body | Baseline
  The Dual-energy X-ray Absorptiometry (DXA) measures the bone mineral density (BMD) of the spine, hip and whole-body.
Bone Mineral Density of Spine, Hip and Whole-body | 2 years
  The Dual-energy X-ray Absorptiometry (DXA) measures the bone mineral density (BMD) of the spine, hip and whole-body.
Bone Area of Spine, Hip and Whole-body | Baseline
  The Dual-energy X-ray Absorptiometry (DXA) measures the bone area (BA) of the spine, hip and whole-body.
Bone Area of Spine, Hip and Whole-body | 2 years
  The Dual-energy X-ray Absorptiometry (DXA) measures the bone area (BA) of the spine, hip and whole-body.
Bone Mineral Content of Spine, Hip and Whole-body | Baseline
  The Dual-energy X-ray Absorptiometry (DXA) measures the bone mineral content (BMC) in the spine, hip and whole-body.
Bone Mineral Content of Spine, Hip and Whole-body | 2 years
  The Dual-energy X-ray Absorptiometry (DXA) measures the bone mineral content (BMC) in the spine, hip and whole-body.

SECONDARY OUTCOMES:
Total Body Lean Mass | Baseline
  The Dual-energy X-ray Absorptiometry (DXA) measures the whole-body densitometry, providing information on total body lean mass in kg.
Total Body Lean Mass | 2 years
  The Dual-energy X-ray Absorptiometry (DXA) measures the whole-body densitometry, providing information on total body lean mass in kg.
Total Body Fat Mass | Baseline
  The Dual-energy X-ray Absorptiometry (DXA) measures the whole-body densitometry, providing information on total body fat mass in kg.
Total Body Fat Mass | 2 years
  The Dual-energy X-ray Absorptiometry (DXA) measures the whole-body densitometry, providing information on total body fat mass in kg.
High-Resolution Peripheral Quantitative Computed Tomography of The Distal Radius and Tibia | Baseline
  High-resolution peripheral quantitative computed tomography (HRpQCT) of the distal radius and tibia will provide structural information including cortical thickness, trabecular number, trabecular thickness and volumetric bone mineral density (vBMD)
High-Resolution Peripheral Quantitative Computed Tomography of The Distal Radius and Tibia | 2 years
  High-resolution peripheral quantitative computed tomography (HRpQCT) of the distal radius and tibia will provide structural information including cortical thickness, trabecular number, trabecular thickness and volumetric bone mineral density (vBMD)
Body Weight | Baseline
  Weight will be measured to the nearest 0.1 kg on an electronic scale with participants wearing light clothing. Measurement will be carried out barefoot.
Body Weight | 2 years
  Weight will be measured to the nearest 0.1 kg on an electronic scale with participants wearing light clothing. Measurement will be carried out barefoot.
Height | Baseline
  Height will be measured to the nearest 0.5 cm using a portable stadiometer. Measurement will be carried out barefoot
Height | 2 years
  Height will be measured to the nearest 0.5 cm using a portable stadiometer. Measurement will be carried out barefoot
Body Mass Index | Baseline
  Body Mass Index (BMI) will be calculated based on the participant's weight and height
Body Mass Index | 2 years
  Body Mass Index (BMI) will be calculated based on the participant's weight and height
Waist Circumference | Baseline
  The waist circumference will be measured using a measuring tape to the nearest 0.5 cm. At least two measurements will be performed and a third will be made if the two differs by more than 1 cm
Waist Circumference | 2 years
  The waist circumference will be measured using a measuring tape to the nearest 0.5 cm. At least two measurements will be performed and a third will be made if the two differs by more than 1 cm
Hip Circumference | Baseline
  The hip circumference will be measured using a measuring tape to the nearest 0.5 cm. At least two measurements will be performed and a third will be made if the two differs by more than 1 cm
Hip Circumference | 2 years
  The hip circumference will be measured using a measuring tape to the nearest 0.5 cm. At least two measurements will be performed and a third will be made if the two differs by more than 1 cm
Waist-Hip Ratio | Baseline
  The waist-hip ratio is calculated using the waist and hip circumference
Waist-Hip Ratio | 2 years
  The waist-hip ratio is calculated using the waist and hip circumference
Endocrine Status | Baseline
  Blood will be drawn for plasma analyses for endocrine status
Endocrine Status and Bone Markers of Bone Metabolism | Baseline
  Blood will be drawn for plasma analyses for endocrine status and biomarkers of bone metabolism (PINP and CTX)
Hair Cortisol Concentrations | Baseline
  The hair samples will be cut from the posterior apex as close to the scalp as possible (minimum 20 mg per participant). Cortisol extracted from the hair will be analysed via the Elisa method
Blood Pressure | Baseline
  Resting blood pressure will be measured
Blood Pressure | 2 years
  Resting blood pressure will be measured

OTHER OUTCOMES:
Self-reported Stress | Baseline
  Information about well-being will be collected by electronic questionnaire, using the World Health Organization Well-Being index (WHO-5): (1) 'I have felt cheerful and in good spirits', (2) 'I have felt calm and relaxed', (3) 'I have felt active and vigorous', (4) 'I woke up feeling fresh and rested' and (5) 'My daily life has been filled with things that interest me'. The respondent is asked to rate how well each of the 5 statements applies to him or her when considering the last 14 days. Each of the 5 items is scored from 5 (all of the time) to 0 (none of the time). Score ranges from 0 (absence of well-being) to 25 (maximal well-being).
Self-reported Sleep | Baseline
  Information about sleep will be collected by electronic questionnaire. The respondent is asked about what time he or she goes to sleep and wakes up on the weekdays and weekends/holidays, as well as five elaborating questions about their sleeping pattern: (1) 'How often do you have poor or restless sleep?', (2) 'How often do you have trouble falling asleep?', (3) 'How often do you wake up too early in the morning?', (4) 'How often do you wake up multiple times at night and have trouble falling asleep again?' and (5) 'Do you snore loudly when you sleep?'. Each of the 5 items is scored from 4 (every day or almost every day) to 1 (rarely or never).
Self-reported Hearing | Baseline
  Information about tinnitus will be collected by electronic questionnaire. The respondent is asked the following five questions: (1) 'After listening to loud music or other sounds/noise, have you then heard any form of sounds in your head or ears, even after turning off the loud music or noise?', (2) 'Do you ever experience sounds in your head or ears without listening to loud music or other sounds first?', (3) 'Are you experiencing it today?', (4) 'Does the sound bother you?' and (5) 'How worried are you that sound can harm your hearing?'. The questions 1 to 3 are answered as yes or no. Question 4 is answered as not bothered; a little bothered or very bothered. Question 5 is I am not concerned; I am a little concerned or I am seriously concerned.

CONTACTS AND LOCATIONS:
Overall Officials: Bo Abrahamsen, MD, PhD, Study Chair — OPEN, University of Southern Denmark, Odense and Department of Medicine 1, Holbæk Hospital, Holbæk; Katrine H Rubin, MHS, PhD, Principal Investigator — OPEN, Department of Clinical Research, University of Southern Denmark and Odense University Hospital; Bente Langdahl, MD, PhD, Principal Investigator — Department of Clinical Medicine and Department of Endocrinology and Diabetes, Aarhus University; Peter Vestergaard, MD, PhD, Principal Investigator — Faculty of Medicine, Aalborg University and Department of Endocrinology, Aalborg University Hospital; Berit L Heitmann, DMD, PhD, Principal Investigator — The Parker Institute, Frederiksberg Hospital, Frederiksberg; Mina N Händel, Msc, PhD, Principal Investigator — The Parker Institute, Frederiksberg Hospital, Frederiksberg; Charlotte L Tofteng, MD, PhD, Principal Investigator — Department of CIinical Medicine, Endocrinology, Zealand University Hospital, Køge; Pernille Bach-Mortensen, MD, PhD, Principal Investigator — Department of Endocrinology, Amager and Hvidovre Hospital, Hvidovre; Pernille Hermann, MD, PhD, Principal Investigator — Department of Endocrinology, Odense University Hospital, Odense; Niklas R Jørgensen, MD, PhD, Principal Investigator — Department of Clinical Biochemistry and Centre of Diagnostic Investigation,Rigshospitalet Copenhagen; Jonas Bybjerg-Grauholm, MSE, Principal Investigator — Danish Center for Neonatal Screening, Statens Serum Institut, Copenhagen
Locations (9):
- Denmark (9):
  - Aalborg University Hospital, Department of Endocrinology, Aalborg
  - Aarhus University Hospital, Department of Endocrinology, Aarhus
  - Rigshospitalet, Department of Clinical Biochemistry and Endocrinology, Copenhagen
  - Bispebjerg and Frederiksberg Hospital, EEK, Parker Institute, Frederiksberg
  - Holbæk Hospital, Department of Medicine, Holbæk
  - Hvidovre Hospital, Department of Endocrinology, Hvidovre
  - Zealand University Hospital, Department of Medicine, Køge
  - Odense University Hospital, Department of Endocrinology, Odense
  - University of Southern Denmark, Department of Clinical Research, Odense

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Yu XH, Wei YY, Zeng P, Lei SF. Birth weight is positively associated with adult osteoporosis risk: observational and Mendelian randomization studies. J Bone Miner Res. 2021 Aug;36(8):1469-1480. doi: 10.1002/jbmr.4316. Epub 2021 Jun 9. PMID 34105796
- [Background] Curtis EM, Fuggle NR, Cooper C, Harvey NC. Epigenetic regulation of bone mass. Best Pract Res Clin Endocrinol Metab. 2022 Mar;36(2):101612. doi: 10.1016/j.beem.2021.101612. Epub 2022 Jan 4. PMID 35120798
- [Background] Krstic N, Bishop N, Curtis B, Cooper C, Harvey N, Lilycrop K, Murray R, Owen R, Reilly G, Skerry T, Borg S. Early life vitamin D depletion and mechanical loading determine methylation changes in the RUNX2, RXRA, and osterix promoters in mice. Genes Nutr. 2022 May 26;17(1):7. doi: 10.1186/s12263-022-00711-0. PMID 35619053
- [Background] Reppe S, Lien TG, Hsu YH, Gautvik VT, Olstad OK, Yu R, Bakke HG, Lyle R, Kringen MK, Glad IK, Gautvik KM. Distinct DNA methylation profiles in bone and blood of osteoporotic and healthy postmenopausal women. Epigenetics. 2017 Aug;12(8):674-687. doi: 10.1080/15592294.2017.1345832. Epub 2017 Jun 26. PMID 28650214
- [Background] Williams GR, Bassett JHD. Thyroid diseases and bone health. J Endocrinol Invest. 2018 Jan;41(1):99-109. doi: 10.1007/s40618-017-0753-4. Epub 2017 Aug 29. PMID 28853052
- [Background] Cardoso I, Specht IO, Thorsteinsdottir F, Thorbek MJ, Keller A, Stougaard M, Cohen AS, Handel MN, Kristensen LE, Heitmann BL. Vitamin D Concentrations at Birth and the Risk of Rheumatoid Arthritis in Early Adulthood: A Danish Population-Based Case-Cohort Study. Nutrients. 2022 Jan 20;14(3):447. doi: 10.3390/nu14030447. PMID 35276806
- [Background] Handel MN, Frederiksen P, Cohen A, Cooper C, Heitmann BL, Abrahamsen B. Neonatal vitamin D status from archived dried blood spots and future risk of fractures in childhood: results from the D-tect study, a population-based case-cohort study. Am J Clin Nutr. 2017 Jul;106(1):155-161. doi: 10.3945/ajcn.116.145599. Epub 2017 May 17. PMID 28515065
- [Background] Jensen CB, Lundqvist M, Sorensen TIA, Heitmann BL. Neonatal Vitamin D Levels in Relation to Risk of Overweight at 7 Years in the Danish D-Tect Case-Cohort Study. Obes Facts. 2017;10(3):273-283. doi: 10.1159/000471881. Epub 2017 Jun 10. PMID 28601865
- [Background] Keller A, Thorsteinsdottir F, Stougaard M, Cardoso I, Frederiksen P, Cohen AS, Vaag A, Jacobsen R, Heitmann BL. Vitamin D concentrations from neonatal dried blood spots and the risk of early-onset type 2 diabetes in the Danish D-tect case-cohort study. Diabetologia. 2021 Jul;64(7):1572-1582. doi: 10.1007/s00125-021-05450-2. Epub 2021 May 24. PMID 34028586
- [Background] Keller A, Frederiksen P, Handel MN, Jacobsen R, McGrath JJ, Cohen AS, Heitmann BL. Environmental and individual predictors of 25-hydroxyvitamin D concentrations in Denmark measured from neonatal dried blood spots: the D-tect study. Br J Nutr. 2019 Mar 14;121(5):567-575. doi: 10.1017/S0007114518003604. Epub 2019 Jan 30. PMID 30526709
- [Background] Keller A, Handel MN, Frederiksen P, Jacobsen R, Cohen AS, McGrath JJ, Heitmann BL. Concentration of 25-hydroxyvitamin D from neonatal dried blood spots and the relation to gestational age, birth weight and Ponderal Index: the D-tect study. Br J Nutr. 2018 Jun;119(12):1416-1423. doi: 10.1017/S0007114518000879. Epub 2018 Apr 25. PMID 29690937
- [Background] Thorsteinsdottir F, Cardoso I, Keller A, Stougaard M, Frederiksen P, Cohen AS, Maslova E, Jacobsen R, Backer V, Heitmann BL. Neonatal Vitamin D Status and Risk of Asthma in Childhood: Results from the D-Tect Study. Nutrients. 2020 Mar 21;12(3):842. doi: 10.3390/nu12030842. PMID 32245170
- [Background] Dugue PA, English DR, MacInnis RJ, Jung CH, Bassett JK, FitzGerald LM, Wong EM, Joo JE, Hopper JL, Southey MC, Giles GG, Milne RL. Reliability of DNA methylation measures from dried blood spots and mononuclear cells using the HumanMethylation450k BeadArray. Sci Rep. 2016 Jul 26;6:30317. doi: 10.1038/srep30317. PMID 27457678
- [Background] Staunstrup NH, Starnawska A, Nyegaard M, Christiansen L, Nielsen AL, Borglum A, Mors O. Genome-wide DNA methylation profiling with MeDIP-seq using archived dried blood spots. Clin Epigenetics. 2016 Jul 26;8:81. doi: 10.1186/s13148-016-0242-1. eCollection 2016. PMID 27462375
- [Background] Ghantous A, Saffery R, Cros MP, Ponsonby AL, Hirschfeld S, Kasten C, Dwyer T, Herceg Z, Hernandez-Vargas H. Optimized DNA extraction from neonatal dried blood spots: application in methylome profiling. BMC Biotechnol. 2014 Jul 1;14:60. doi: 10.1186/1472-6750-14-60. PMID 24980254
- [Background] Weaver CM, Gordon CM, Janz KF, Kalkwarf HJ, Lappe JM, Lewis R, O'Karma M, Wallace TC, Zemel BS. The National Osteoporosis Foundation's position statement on peak bone mass development and lifestyle factors: a systematic review and implementation recommendations. Osteoporos Int. 2016 Apr;27(4):1281-1386. doi: 10.1007/s00198-015-3440-3. Epub 2016 Feb 8. PMID 26856587
- [Background] Hannon E, Schendel D, Ladd-Acosta C, Grove J, Hansen CS, Hougaard DM, Bresnahan M, Mors O, Hollegaard MV, Baekvad-Hansen M, Hornig M, Mortensen PB, Borglum AD, Werge T, Pedersen MG, Nordentoft M; iPSYCH-Broad ASD Group; Buxbaum JD, Daniele Fallin M, Bybjerg-Grauholm J, Reichenberg A, Mill J. Variable DNA methylation in neonates mediates the association between prenatal smoking and birth weight. Philos Trans R Soc Lond B Biol Sci. 2019 Apr 15;374(1770):20180120. doi: 10.1098/rstb.2018.0120. PMID 30966880
- [Background] Gicquel C, El-Osta A, Le Bouc Y. Epigenetic regulation and fetal programming. Best Pract Res Clin Endocrinol Metab. 2008 Feb;22(1):1-16. doi: 10.1016/j.beem.2007.07.009. PMID 18279777
- [Background] Jensen KH, Riis KR, Abrahamsen B, Handel MN. Nutrients, Diet, and Other Factors in Prenatal Life and Bone Health in Young Adults: A Systematic Review of Longitudinal Studies. Nutrients. 2020 Sep 19;12(9):2866. doi: 10.3390/nu12092866. PMID 32961712
- [Background] Harvey N, Dennison E, Cooper C. Osteoporosis: a lifecourse approach. J Bone Miner Res. 2014 Sep;29(9):1917-25. doi: 10.1002/jbmr.2286. PMID 24861883
- [Background] Gluckman PD, Hanson MA, Cooper C, Thornburg KL. Effect of in utero and early-life conditions on adult health and disease. N Engl J Med. 2008 Jul 3;359(1):61-73. doi: 10.1056/NEJMra0708473. No abstract available. PMID 18596274
- [Background] Lillycrop K, Murray R, Cheong C, Teh AL, Clarke-Harris R, Barton S, Costello P, Garratt E, Cook E, Titcombe P, Shunmuganathan B, Liew SJ, Chua YC, Lin X, Wu Y, Burdge GC, Cooper C, Inskip HM, Karnani N, Hopkins JC, Childs CE, Chavez CP, Calder PC, Yap F, Lee YS, Chong YS, Melton PE, Beilin L, Huang RC, Gluckman PD, Harvey N, Hanson MA, Holbrook JD; EpiGen Consortium; Godfrey KM. ANRIL Promoter DNA Methylation: A Perinatal Marker for Later Adiposity. EBioMedicine. 2017 May;19:60-72. doi: 10.1016/j.ebiom.2017.03.037. Epub 2017 Apr 26. PMID 28473239
- [Background] Godfrey KM, Costello PM, Lillycrop KA. The developmental environment, epigenetic biomarkers and long-term health. J Dev Orig Health Dis. 2015 Oct;6(5):399-406. doi: 10.1017/S204017441500121X. Epub 2015 May 28. PMID 26017068
- [Background] Block T, El-Osta A. Epigenetic programming, early life nutrition and the risk of metabolic disease. Atherosclerosis. 2017 Nov;266:31-40. doi: 10.1016/j.atherosclerosis.2017.09.003. Epub 2017 Sep 5. PMID 28950165
- [Background] Godfrey KM, Costello PM, Lillycrop KA. Development, Epigenetics and Metabolic Programming. Nestle Nutr Inst Workshop Ser. 2016;85:71-80. doi: 10.1159/000439488. Epub 2016 Apr 18. PMID 27088334
- [Background] Godfrey KM, Sheppard A, Gluckman PD, Lillycrop KA, Burdge GC, McLean C, Rodford J, Slater-Jefferies JL, Garratt E, Crozier SR, Emerald BS, Gale CR, Inskip HM, Cooper C, Hanson MA. Epigenetic gene promoter methylation at birth is associated with child's later adiposity. Diabetes. 2011 May;60(5):1528-34. doi: 10.2337/db10-0979. Epub 2011 Apr 6. PMID 21471513
- [Background] Godfrey KM, Lillycrop KA, Burdge GC, Gluckman PD, Hanson MA. Epigenetic mechanisms and the mismatch concept of the developmental origins of health and disease. Pediatr Res. 2007 May;61(5 Pt 2):5R-10R. doi: 10.1203/pdr.0b013e318045bedb. PMID 17413851
- [Background] Hollegaard MV, Grauholm J, Norgaard-Pedersen B, Hougaard DM. DNA methylome profiling using neonatal dried blood spot samples: a proof-of-principle study. Mol Genet Metab. 2013 Apr;108(4):225-31. doi: 10.1016/j.ymgme.2013.01.016. Epub 2013 Feb 1. PMID 23422032
- [Derived] Handel MN, Jorgensen NR, Bybjerg-Grauholm J, Jansen RB, Eiken P, Tofteng CL, Hermann AP, Bach-Mortensen P, Heitmann BL, Rubin KH, Langdahl BL, Vestergaard P, Abrahamsen B. Early life determinants of skeletal maturation, body composition and endocrine health in young adults (EPIPEAK): protocol for a nationwide birth cohort study. BMJ Open. 2025 Oct 23;15(10):e101632. doi: 10.1136/bmjopen-2025-101632. PMID 41130671